CLINICAL TRIAL: NCT02085109
Title: The Effects of a Diet Rich in Fat or Theobromine on Intestinal apoA-I mRNA and Protein Expression
Brief Title: The Effects of Fat and Theobromine on apoA-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 13-3-049
Record Dates: First submitted 2014-02-17; First posted 2014-03-12 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; HDL metabolism; ApoA-I; High fat; Theobromine
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Theobromine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High fat meal (Experimental): A high fat milkshake containing 60.6 grams of fat
  Interventions: Dietary Supplement: Fat milkshake
- Low fat meal (Placebo Comparator): A Low fat milkshake containing 10.5 gram of fat
  Interventions: Dietary Supplement: Fat milkshake
- A Low fat meal containing theobromine (Experimental): A low fat milkshake containing 10.5 grams of fat supplemented with 850 mg of theobromine
  Interventions: Dietary Supplement: Fat milkshake; Dietary Supplement: Theobromine

INTERVENTIONS:
Dietary Supplement: Fat milkshake
Dietary Supplement: Theobromine
  Arms: A Low fat meal containing theobromine

SUMMARY:
Rationale: Despite successful efforts to lower atherogenic serum low-density lipoprotein (LDL) cholesterol concentrations, a substantial residual cardiovascular risk is still present. An additive strategy to further lower this residual risk may be via raising high-density lipoprotein (HDL) cholesterol concentrations, and in particular those of its major protein constituent apolipoprotein A-I (apoA-I). However, recent evidence shows that raising HDL cholesterol (HDL-C) concentrations not always causes a reduction in cardiovascular disease (CVD) risk. To understand this it is important to know what are the targets and molecular mechanisms that underlie a shift to a HDL fraction with cardioprotective activities. There is increasing evidence that particularly the apoA-I proteins in the HDL fractions are atheroprotective. It is important to verify whether the effect of an intervention actually increases apoA-I production since that results in the formation of de-novo small pre-beta HDL particles that have full capacity to resorb cholesterol from the arterial wall and return this to the liver for secretion (reverse cholesterol transport). The investigators here propose to evaluate, in a double-blind human intervention study, the difference in intestinal apoA-I gene expression, of healthy subjects, after consumption of a high fat (HF) or low fat (LF) meal. Additionally the investigators propose to evaluate the effect of theobromine on intestinal apoA-I expression. Based on several studies, theobromine improved cardiovascular risk parameters among which an elevation in apoA-I and HDL cholesterol concentrations. It is however unknown whether this effect of theobromine originates from elevated apoA-I production, which suggest improved functionality, or decreased clearance, suggesting reduced functionality. The investigators therefore propose to also evaluate if the usage of theobromine is a better way to increase intestinal apoA-I mRNA and protein expression, than consumption of a HF meal. The investigators will do this in the same double-blind human intervention study. The theobromine will be added in a third arm in a LF condition.

Study design: The proposed study will have a randomized, double-blind cross-over design. The total study duration will be 17 days, consisting of 3 experimental days with postprandial tests, each separated by a 1 week wash-out period.

Study population: Ten apparently healthy male subjects, aged 18-60 years, without a history of any gastrointestinal disorders or complaints.

Intervention: During the three experimental days, subjects will consume a milkshake: one HF milkshake, one LF milkshake and one LF milkshake supplemented with 850 mg theobromine. Total follow-up during each of the postprandial tests is 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years
* Serum total cholesterol <8.0 mmol/L
* Plasma glucose <7.0 mmol/L
* BMI between 20 - 30 kg/m2
* Non-smoking
* Willingness to abstain from theobromine rich products from two weeks prior to the study maintaining throughout the full duration (17 days) of the study:

  * Chocolate containing products (see Appendix A).
* Willingness to abstain from energy drinks from two weeks prior to the study maintaining throughout the full duration (17 days) of the study, because of its high caffeine content,
* Willingness to reduce caffeine containing drinks till maximum 4 drinks a day from two weeks prior to the study maintaining throughout the full duration (17 days) of the study:

  * Coffee
  * Tea
  * Cola.

Exclusion Criteria:

* Unstable body weight (weight gain or loss >3 kg in the past 3 months),
* Not willing to stop the consumption of gastric acid inhibitor, laxantia, prebiotics, probiotics and antibiotics for at least one month before the start of the study and during the study.
* Any medical condition requiring treatment and/or medication use,
* Indication for treatment with cholesterol-lowering drugs according to the Dutch Cholesterol Consensus (35)
* Use of medication or a medically-prescribed diet known to affect serum lipid or glucose metabolism. The use of oral contraceptives and paracetamol is allowed.
* Active cardiovascular disease (for instance congestive heart failure) or recent (<6 months) event, such as acute myocardial infarction or cerebro-vascular accident.
* Gastrointestinal diseases (like celiac disease, inflammatory bowel disease, irritable bowel disease and food allergies) or a history of any gastrointestinal disorders or complaints.
* Severe medical conditions that might interfere with the study such as epilepsy, asthma, chronic obstructive pulmonary disease and rheumatoid arthritis.
* Not willing to stop the consumption of vitamin supplements or fish oil capsules 3 weeks before the start of the study
* Consumption of >21 glasses of alcohol-containing drinks per week.
* Abuse of drugs
* Participation in another biomedical study within 1 month prior to the screening visit
* Having donated > 150 ml blood within 1 month prior to the screening visit, planning to donate blood during the study or within one month after finishing the study.
* Impossible or difficult to puncture as evidenced during the screening visits.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Microarray | up to 3 days
  On each 3 test days 5 hours after the postprandial meal a biopsy will be taken. From these intestinal cells gene expression profiles will be measured by microarray.

SECONDARY OUTCOMES:
Blood samples | Day 1, 2 and 3 at T=0, 15, 30, 45, 60, 90, 120, 180 and 240 min
  During each test day blood samples will be taken in intervals after consumption of the postprandial meal. Blood samples are taken to analyse lipids, apoA-I, apoB-100, apoB48, CRP, cholesterol efflux, glucose and free fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Prof, Principal Investigator — Maastricht University Hospital; Ronald Mensink, Prof, Study Director — Maastricht University Hospital
Locations (1):
- Maastricht University Hospital, Maastricht, Netherlands